CLINICAL TRIAL: NCT06577311
Title: An Investigator Initiated Study to Evaluate the Safety and Efficacy of Aminolevulinic Acid Hydrochloride Topical Gel, 10% (Ameluz ®) With RhodoLED-XL® Red Light in the Treatment of Facial Cutaneous Squamous Cell Carcinoma in Situ (SCCis)"
Brief Title: Evaluating the Use of Photodynamic Therapy to Treat Facial Cutaneous Squamous Cell Carcinoma in Situ (SCCis)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: Biofrontera Inc. (Industry)
Responsible Party: Principal Investigator, Mark Steven Nestor, M.D., Ph.D., Director, The Center for Clinical and Cosmetic Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCR 01-2024
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: skin cancer; facial skin cancer; Squamous Cell Carcinoma; Squamous Cell Carcinoma in Situ; Cutaneous Squamous Cell Carcinoma in Situ; Facial Cutaneous Squamous Cell Carcinoma in Situ; SCCis
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Squamous Cell; Squamous Intraepithelial Lesions | interventions — Aminolevulinic Acid; Gels; Red Light

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Photodynamic Therapy (using Red light dose) (Experimental): 20 participants will be enrolled to this arm
  Interventions: Combination Product: Aminolevulinic acid hydrochloride 10% topical gel with Red Light

INTERVENTIONS:
Combination Product: Aminolevulinic acid hydrochloride 10% topical gel with Red Light — Participants will have their facial Cutaneous Squamous Cell Carcinoma in situ (SCCis) prepped then treated with Aminolevulinic acid hydrochloride 10% topical gel (Ameluz ®), followed by red light therapy administered for 13 minutes and 30 seconds to deliver the total desired light dose to the SCCis lesion.
  Other Names: Ameluz ®; RhodoLED-XL®

SUMMARY:
The goal of this clinical trial is to test how safe and effective it is to treat early form of cancer cells found in the upper skin layer of the face, using a light-sensitive gel used in combination with a light source.

The main questions this trial aims to answer are:

* to confirm using laboratory testing, how much of the affected facial skin cancer section the treatment was able to remove, and;
* seeing how many participants had no remaining affected facial skin cancer sections after treatment.

Participants who qualify will be asked to complete 14 visits in total and will receive a total of two treatments, after voluntarily consent has been given.

DETAILED DESCRIPTION:
In the study, participants will be asked to complete the following:

* Provide basic personal information (including date of birth, gender, race and ethnicity)
* Provide their medical/ surgical history and perform a medical exam (including but not limited to symptom-directed physical exam, skin type, vital signs, height, weight and urine pregnancy test collection)
* Follow study rules such as avoiding certain medications and treatments
* Provide information on any medications, treatments or reactions that started after the study began
* Allow two treatments on the skin cancer area of the face using a light-sensitive cream used in combination with a light source
* Allow clinical documentation of the treatment, such as how well the treatment was tolerated, any skin reaction or side effects
* Allow surgery to remove the skin cancer area from the face for Laboratory testing

To qualify for this trial, participants must:

* be an adult (18 years of age or older)
* give voluntary written consent
* have a recently diagnosed (less than six months from first visit) skin cancer area on the face that meets surgery size requirements
* be willing to follow study instructions and complete study requirements, including not using non-approved lotions and creams on the treatments areas
* allow photographs of the area of skin cancer being treated on the face
* (if female) not be pregnant before and during the study and agree to use acceptable forms of birth control
* confirm they are not sensitive to any of the study treatment ingredients

All surgery samples collected from the participants towards the end of the study will be sent to a laboratory for testing. All photographs of the treatment area collected during the study will be used as study data.

All participants have the right to refuse further participation in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Must be an adult (18 years of age or older)
* Must have a recently diagnosed (no more than six months from first study visit) facial SCCis lesion that meets surgery excision size requirements
* Cannot have other dermatological disease in the SCCis target area
* Must be willing to follow study instructions and complete study requirements, including not using non-approved lotions and creams on the treatments areas
* Voluntary written consent required
* Allow photographs of the area of skin cancer being treated on the face
* Agree to use acceptable forms of birth control. If female, cannot be pregnant before and during the study

Exclusion Criteria:

* Pregnant or lactating
* Sensitive to any of the study treatment ingredients
* Medical laboratory evidence of other non-SCCis tumor in the target lesion biopsy specimen
* History of recurrence if the target SCCis lesion
* Evidence of dermatological disease or skin condition in the treatment area
* Medical laboratory evidence of growth patterns in the target lesion biopsy specimen
* Chronic medical condition that in the Investigators opinion will interfere in the trial or affect participant safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with histological clearance of treated SCCis lesion. | an average of 12 weeks
  Histological clearance is defined as the absence of detectable evidence of SCCis tumor cell nests by the central pathology reports

SECONDARY OUTCOMES:
Number of participants with clinical clearance of treated SCCis lesion | an average of 12 weeks
  Complete Clinical Clearance will be measured by the Investigator and is defined as when there is no clinically visible lesion remaining at the site
Size of the lesion | Up to 16 weeks
  Changes noted in the size of the treated SCCis lesion site, measured by the longest diameter.
Local Skin Response Scale | Up to 16 weeks
  Observations and changes noted in the aesthetic appearance (Erythema, Flaking/Scaling, Crusting, Swelling, Vesiculation/ Pustulation, Erosion/ Ulceration) of thetreated isSCC lesion will each be graded on a scale of 0 to 4, with 0 as no presenceand 4 as a severe outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, MD, PhD, Principal Investigator — Center for Clinical and Cosmetic Research
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States